CLINICAL TRIAL: NCT03782792
Title: Effisayil™ 1:Multi-center, Double-blind, Randomised, Placebo-controlled, Phase II Study to Evaluate Efficacy, Safety and Tolerability of a Single Intravenous Dose of Spesolimab (BI 655130) in Patients With Generalized Pustular Psoriasis (GPP) Presenting With an Acute Flare of Moderate to Severe Intensity
Brief Title: Effisayil™ 1: A Study to Test Spesolimab (BI 655130) in Patients With a Flare-up of a Skin Disease Called Generalized Pustular Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0013; 2017-004231-37 (EudraCT Number)
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spesolimab — Solution for infusion
  Other Names: BI 655130
  Arms: Spesolimab
Drug: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
To evaluate efficacy, safety, and tolerability of spesolimab (BI 655130) compared to placebo in patients with Generalized Pustular Psoriasis (GPP) presenting with an acute flare of moderate to severe intensity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GPPGA of 0 or 1 and a known and documented history of GPP per European Rare And Severe Psoriasis Expert Network (ERASPEN) criteria regardless of IL36RN mutation status, with previous evidence of fever, and/or asthenia, and/or myalgia, and/or elevated C-reactive protein, and/or leucocytosis with peripheral blood neutrophilia (above ULN) OR

  -- Patients with an acute flare of moderate to severe intensity meeting the (ERASPEN) criteria of GPP with a known and documented history of GPP (per ERASPEN criteria) regardless of IL36RN mutation status, with previous evidence of fever, and/or asthenia, and/or myalgia, and/or elevated C-reactive protein, and/or leucocytosis with peripheral blood neutrophilia (above ULN)
* Male or female patients, aged 18 to 75 years at screening.
* Signed and dated written informed consent prior to admission to the study in accordance with ICH GCP and local legislation prior to start of any screening procedures.
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. Note: A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is not a method of permanent sterilization. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause
* Further inclusion criteria apply

Exclusion Criteria:

* Patients with SAPHO (Synovitis-acne-pustulosis-hyperostosis-osteitis) syndrome.
* Patients with primary erythrodermic psoriasis vulgaris.
* Patients with primary plaque psoriasis vulgaris without presence of pustules or with pustules that are restricted to psoriatic plaques.
* Drug-triggered Acute Generalized Exanthematous Pustulosis (AGEP).
* Immediate life-threatening flare of GPP or requiring intensive care treatment, according to the investigator's judgement. Life-threatening complications mainly include, but are not limited to, cardiovascular/cytokine driven shock, pulmonary distress syndrome, or renal failure.
* Severe, progressive, or uncontrolled hepatic disease, defined as >3- fold Upper Limit of Normal (ULN) elevation in AST or ALT or alkaline phosphatase, or >2-fold ULN elevation in total bilirubin.
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
- China (5):
  - The First Hospital of Dalian Medical University, Dalian
  - 2nd Affiliated Hosp Zhejiang University College of Medical, Hangzhou
  - Shanghai Skin Disease Hospital, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
- France (3):
  - HOP Saint-André, Bordeaux
  - HOP Saint-Louis, Paris
  - HOP Robert Debré, Reims
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Essen AöR, Essen
  - Klinikum der Universität München - Campus Innenstadt, München
- Japan (6):
  - Nagoya City University Hospital, Aichi, Nagoya
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Asahikawa Medical University Hospital, Hokkaido, Asahikawa
  - Tohoku University Hospital, Miyagi, Sendai
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
- Malaysia (7):
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Selayang, Kuala Selangor
  - Hospital Pakar Sultanah Fatimah, Muar town
  - Hospital Raja Permaisuri Bainun, Negeri Perak/Ipoh
  - Hospital Pulau Pinang, Pulau Pinang
- National University Hospital, Singapore, Singapore
- Severance Hospital, Seoul, South Korea
- University Hospital of Lausanne, Lausanne, Switzerland
- National Taiwan University Hospital, Taipei, Taiwan
- Ramathibodi Hospital, Ratchatewi, Bangkok, Thailand
- Tunisia (3):
  - Farhat Hached Hospital, Sousse
  - La Rabta Hospital, Tunis
  - Hedi Chaker Hospital, Department of Dermatology, Tunisia

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- [Derived] Gwillim EC, Nichols AJ. Spesolimab for generalized pustular psoriasis: a review of two key clinical trials supporting initial US regulatory approval. Front Immunol. 2024 Jul 22;15:1359481. doi: 10.3389/fimmu.2024.1359481. eCollection 2024. PMID 39104539
- [Derived] Tsai TF, Zheng M, Ding Y, Song Z, Liu Q, Chen Y, Hu H, Xu J. Efficacy and Safety of Spesolimab in Patients with Generalized Pustular Psoriasis: A Subgroup Analysis of Chinese Patients in the Effisayil 1 Trial. Dermatol Ther (Heidelb). 2023 Dec;13(12):3097-3110. doi: 10.1007/s13555-023-01037-4. Epub 2023 Oct 16. PMID 37840119
- [Derived] Bachelez H, Choon SE, Marrakchi S, Burden AD, Tsai TF, Morita A, Navarini AA, Zheng M, Xu J, Turki H, Anadkat MJ, Rajeswari S, Hua H, Vulcu SD, Hall D, Tetzlaff K, Thoma C, Lebwohl MG; Effisayil 1 Trial Investigators. Trial of Spesolimab for Generalized Pustular Psoriasis. N Engl J Med. 2021 Dec 23;385(26):2431-2440. doi: 10.1056/NEJMoa2111563. PMID 34936739
- [Derived] Choon SE, Lebwohl MG, Marrakchi S, Burden AD, Tsai TF, Morita A, Navarini AA, Zheng M, Xu J, Turki H, Rajeswari S, Deng H, Tetzlaff K, Thoma C, Bachelez H. Study protocol of the global Effisayil 1 Phase II, multicentre, randomised, double-blind, placebo-controlled trial of spesolimab in patients with generalized pustular psoriasis presenting with an acute flare. BMJ Open. 2021 Mar 30;11(3):e043666. doi: 10.1136/bmjopen-2020-043666. PMID 33785490
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, double-blind, parallel-group, single-dose trial with 2 treatment groups (spesolimab and placebo) to evaluate efficacy, tolerability, and safety of spesolimab (BI 655130) compared with placebo in patients with Generalized Pustular Psoriasis (GPP) presenting with an acute flare of moderate to severe intensity.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Patients received intravenously (i.v.) solution for infusion containing 900 milligram (mg) of placebo to spesolimab on Day 1 (D1) of Week 1 (Wk1). Based on the subsequent treatment response, participants were then to be followed up for 12 to 28 weeks. If the severity and progression of the disease worsened within the first week the investigator could treat the patient with a Standard of Care (SoC) treatment of his/her choice (escape medication). If the disease condition was stable, it was recommended to wait until the primary endpoint visit (Wk1/D8) before prescribing an escape medication (SoC) since there was an option to administer open label (OL) spesolimab instead at this time. If escape medication was administered within the first week, the patient was not eligible to receive treatment with a single OL i.v. dose of 900 mg spesolimab on D8. If the condition of the patients worsened after Wk1/D8 patients were eligible to receive rescue treatment with open label spesolimab (only one single rescue i.v. dose of 900 mg spesolimab) after Wk1 to Wk 12.
- Spesolimab 900 mg i.v SD: Patients received intravenously (i.v.) a single dose (SD) of solution for infusion containing 900 milligram (mg) of spesolimab on Day 1 (D1) of Week 1 (Wk1). Based on the subsequent treatment response, participants were then to be followed up for 12 to 28 weeks.
  If the severity and progression of the disease worsened within the first week the investigator could treat the patient with a Standard of Care (SoC) treatment of his/her choice (escape medication). If the disease condition was stable, it was recommended to wait until the primary endpoint visit (Wk1/D8) before prescribing an escape medication (SoC) since there was an option to administer open label (OL) spesolimab instead at this time. If escape medication was administered within the first week, the patient was not eligible to receive treatment with a single OL i.v. dose of 900 mg spesolimab on D8.
  If the condition of the patients worsened after Wk1/D8 patients were eligible to receive rescue treatment with open label spesolimab (only one single rescue i.v. dose of 900 mg spesolimab) after Wk1 to Wk 12.
Period: Overall Study
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Started | 18 | 35
Received Open Label Treatment With Spesolimab at Wk1/D8 (In addition to the randomized treatment, patients received also an i.v. dose of 900 mg spesolimab at Wk1/D8.) | 15 | 12
Received Rescue Treatment With Spesolimab After Wk1 (In addition to the randomized treatment, Patients received also one single rescue i.v. dose of 900 mg spesolimab between Wk1 to Wk 12.) | 2 | 4
Completed (Completed planned observation period.) | 17 | 32
Not Completed | 1 | 3
Not completed — Patient left the country | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS): This patient set included all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spesolimab 900 mg i.v SD | Total
Number analyzed (Participants) | 18 | 35 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.6 (8.4) | 43.2 (12.1) | 43.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 3 | 14 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 35 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 16 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 19 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) Pustulation Subscore of 0 Indicating no Visible Pustules at Week 1
Description: The Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) relies on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The investigator (or qualified site personnel) scored the erythema, pustules, and scaling of all GPP lesions from 0 to 4.
  The GPPGA pustulation subscore ranges from 0 to 4 where:
  0 = clear;
  1. = almost clear;
  2. = mild:
  3. = moderate;
  4. = severe. A lower GPPGA pustulation subscore indicates a better outcome. A GPPGA pustulation subscore of 0 means no visible pustules.
  The proportion of patients who achieved a GPPGA pustulation subscore of 0 at Week 1 is reported.
Time Frame: At Week 1.
Population: Randomized Set (RS) (via estimand EN-NRI): This patient set included all randomized patients. EN = Any assessments after death, or any use of escape medication due to disease worsening (defined as worsening of clinical status or GPP skin and/or systemic symptoms as defined by the investigator) prior to Week 1 were considered to represent a non-response. NRI = Non-response imputation for any missing data.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.056 [0.010 to 0.258] | 0.543 [0.382 to 0.695]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; The Suissa-Shuster Z-pooled test was implemented to test the treatment effect on the primary endpoint on the RS (estimand EN) at a 1-sided, alpha level of 0.025. Confidence intervals (95%) around the risk difference were produced using the Chan and Zhang method; Test type: Other; p = 0.0004, Suissa-Shuster Z-pooled test — One-sided P Value; Risk Difference (RD) = 0.487, 95% CI 2-sided [0.215 to 0.672] — Risk difference=Response rate of spesolimab - response rate of placebo

2. Secondary Outcome: Key Secondary: Proportion of Patients With a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) Score of 0 or 1 at Week 1
Description: GPPGA relied on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The GPPGA total score was calculated by taking the mean of the erythema subscore, pustules subscore and scaling/crusting subscore. The severity of each subscore was assessed using a 5 point scale score ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). The final GPPGA score is assigned as follows:
  * 0, if scores for all three subscores are 0,
  * 1, if 0 < mean < 1.5,
  * 2, if 1.5 ≤ mean < 2.5,
  * 3, if 2.5 ≤ mean < 3.5,
  * 4, if mean ≥ 3.5. A lower GPPGA score indicates a better outcome, with 0 being clear and 1 being almost clear. The proportion of patients with a GPPGA score of 0 or 1 at Week 1 is reported.
Time Frame: At Week 1.
Population: Randomized Set (RS) (via estimand EN-NRI): This patient set included all randomized patients. EN =Any assessments after death, or any use of escape medication due to disease worsening (defined as worsening of clinical status or GPP skin and/or systemic symptoms as defined by the investigator) prior to Week 1 were considered to represent a non-response. NRI = Non-response imputation for any missing data.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.111 [0.031 to 0.328] | 0.429 [0.280 to 0.591]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; The Suissa-Shuster Z-pooled test was implemented to test the treatment effect on the RS (estimand EN) at a 1-sided, alpha level of 0.025. Confidence intervals (95%) around the risk difference were produced using the Chan and Zhang method; Test type: Other; p = 0.0118, Suissa-Shuster Z-pooled test — One-sided P Value; Risk Difference (RD) = 0.317, 95% CI 2-sided [0.022 to 0.527] — Risk difference=Response rate of spesolimab - response rate of placebo

3. Secondary Outcome: Proportion of Patients With a Psoriasis Area and Severity Index for Generalized Pustular Psoriasis (GPPASI) 75 at Week 4
Description: Generalized Pustular Psoriasis Area and Severity Index (GPPASI) provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs).
  A higher score indicates a worse disease state, while a score of 0 indicates no disease. GPPASI 75 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 75% reduction.
  Proportion of patients with GPPASI 75 at Week 4 is reported.
Time Frame: At Week 4.
Population: Randomized Set (RS) (via estimand EN-NRI): This patient set included all randomized patients. EN = Any assessments after death, or any use of escape medication before or after Day 8, open-label spesolimab at Day 8, or rescue medication with spesolimab after Day 8 were considered to represent a non-response. NRI = Non-response imputation for any missing data.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.111 [0.031 to 0.328] | 0.457 [0.305 to 0.618]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0081, Suissa-Shuster Z-pooled test — One-sided P Value; Risk Difference (RD) = 0.346, 95% CI 2-sided [0.058 to 0.554] — Risk difference=Response rate of spesolimab - response rate of placebo

4. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (VAS) Score at Week 4
Description: The pain Visual Analogue Scale (VAS) is a participant-administered single-item scale designed to measure skin pain intensity from generalized pustular psoriasis (GPP) using a 100 millimeter (mm) horizontal VAS. Overall severity of participant's skin pain from GPP is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (pain as bad as one can imagine).
  Change from baseline was calculated by subtracting the VAS score at baseline from the VAS score at Week 4. A negative change indicates an improvement from baseline.
  Death, any use of escape medication, OL Spesolimab at Day 8, or rescue medication with Spesolimab after Day 8, prior to observing the endpoint was considered to reflect a failure to achieve the endpoint outcome, i.e. non-response (NR).
  NR is not a missing value but the worst possible outcome of the endpoint. For example, if the achieved data is (NR, NR, NR, NR, NR, NR, 2, 3, 3, 3, 5) then Q1 is NR, median is NR and Q3 is 3.
Time Frame: Baseline and at Week 4.
Population: Randomized Set (RS) (via estimand EN-LOCF): This patient set included all randomized patients. EN = Death or any use of escape medication before or after Day 8, open-label spesolimab at Day 8, or rescue medication with spesolimab after Day 8 were considered to represent a non-response and assigned with the worst possible outcomes in rank analysis. LOCF = last observation carried forward imputation for any missing data.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Units on a scale | NA [NA to NA] — NA = "non-response", the worst possible outcome. | -22.45 [-70.41 to NA] — NA = "non-response", the worst possible outcome.
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; The effect of spesolimab was evaluated by a Wilcoxon rank test using the RS. Any assessments after death, the use of escape medication (before or after Day 8), open label spesolimab on Day 8, or rescue medication with spesolimab after Day 8 were assigned worst ranks for the testing. Missing data at Week 4 were imputed and handled via assessment of ranks; Test type: Other; p = 0.0012, Wilcoxon (Mann-Whitney) — One-sided P Value; The difference between treatments, based on the RS, using a modified Hodges-Lehmann (HL) estimate of the median difference and 95% Confidence Intervals could not be calculated due to lack of valid data

5. Secondary Outcome: Change From Baseline in Psoriasis Symptom Scale (PSS) Score at Week 4
Description: PSS is a 4-item patient-reported outcome instrument that assesses the severity of psoriasis symptoms in moderate to severe psoriasis patients. The symptoms included are: pain, redness, itching, and burning. The symptom severity was assessed using a 5 point scale ranging from 0 to 4 where 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe. The symptom scores are added to an unweighted total score (range: 0 to 16). A lower PSS score indicates a better outcome. Change from baseline =PSS score at Week 4 - PSS score at baseline. Death, any use of escape medication, OL Spesolimab at Day 8, or rescue medication with Spesolimab after Day 8, prior to observing the endpoint was considered to reflect a failure to achieve the endpoint outcome, i.e. non-response (NR). NR is not a missing value but the worst possible outcome of the endpoint. For example, if the achieved data is (NR, NR, NR, NR, NR, NR, 2, 3, 3, 3, 5) then Q1 is NR, median is NR and Q3 is 3.
Time Frame: Baseline and at Week 4.
Population: Randomized Set (RS) (via estimand EN-LOCF): This patient set included all randomized patients. EN = Any assessments after death, or any use of escape medication before or after Day 8, open-label spesolimab at Day 8, or rescue medication with spesolimab after Day 8 were considered to represent a non-response and assigned with the worst possible outcomes in rank analysis. LOCF = last observation carried forward imputation for any missing data.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Units on a scale | NA [NA to NA] — NA = "non-response", the worst possible outcome. | -2.0 [-9.0 to NA] — NA = "non-response", the worst possible outcome.
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0044, Wilcoxon (Mann-Whitney) — One-sided P Value; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Score at Week 4
Description: The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Each items is scored from 0 to 4. Score range is 0 (extreme fatigue)-52 (no fatigue).
  Change from baseline=FACIT Fatigue score at Week 4- FACIT-Fatigue score at baseline. Death, any use of escape medication, OL Spesolimab at Day 8, or rescue medication with Spesolimab after Day 8, prior to observing the endpoint was considered to reflect a failure to achieve the endpoint outcome, i.e. non-response (NR). NR is not a missing value but the worst possible outcome of the endpoint. For example, if the achieved data is s (NR, NR, NR, NR, NR, NR, 2, 3, 3, 3, 5) then Q1 is NR, median is NR and Q3 is 3.
Time Frame: Baseline and at Week 4.
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Units on a scale | NA [NA to NA] — NA = "non-response", the worst possible outcome. | 3.00 [NA to 30.00] — NA = "non-response", the worst possible outcome.
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0012, Wilcoxon (Mann-Whitney) — One-sided P Value; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: Proportion of Patients With a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) Score of 0 or 1 at Week 4
Description: GPPGA relied on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The GPPGA total score is calculated by taking the mean of the erythema subscore, pustules subscore and scaling/crusting subscore. The severity of each subscore was assessed using a 5 point scale score ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). The final GPPGA score is assigned as follows:
  * 0, if scores for all three scores are 0,
  * 1, if 0 < mean < 1.5,
  * 2, if 1.5 ≤ mean < 2.5,
  * 3, if 2.5 ≤ mean < 3.5,
  * 4, if mean ≥ 3.5. A lower GPPGA score indicates a better outcome, with 0 being clear and 1 being almost clear.
  The proportion of participants with a GPPGA score of 0 or 1 at Week 4 is reported.
Time Frame: At Week 4.
Population: Randomized Set (RS) (via estimand EN-NRI): This patient set included all randomized patients. EN = Any assessments after death, or the use of escape medication (before or after Day 8), or open-label spesolimab at Day 8, or rescue medication with spesolimab after Day 8, was considered a failure to achieve the endpoint outcome (i.e. non-response). NRI = Non-response imputation for any missing data.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.111 [0.031 to 0.328] | 0.486 [0.330 to 0.644]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; Confidence intervals (95%) around the risk difference were produced using the Chan and Zhang method; Test type: Other; Risk Difference (RD) = 0.375, 95% CI 2-sided [0.058 to 0.581] — Risk difference=Response rate of spesolimab - response rate of placebo

8. Secondary Outcome: Proportion of Patients With a Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) Pustulation Sub-score of 0 Indicating no Visible Pustules at Week 4
Description: The Generalized Pustular Psoriasis Physician Global Assessment (GPPGA) relies on clinical assessment of the Generalized Pustular Psoriasis (GPP) patient's skin presentation. The investigator (or qualified site personnel) scores the erythema, pustules, and scaling of all GPP lesions from 0 to 4.
  The GPPGA pustulation subscore ranges from 0 to 4 where:
  0 = clear;
  1. = almost clear;
  2. = mild:
  3. = moderate;
  4. = severe. A lower GPPGA pustulation subscore indicates a better outcome. The proportion of patients who achieved a GPPGA pustulation subscore of 0 at Week 1 is reported.
Time Frame: At Week 4.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.111 [0.031 to 0.328] | 0.514 [0.356 to 0.670]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; Confidence intervals (95%) around the risk difference were produced using the Chan and Zhang method; Test type: Other; Risk Difference (RD) = 0.403, 95% CI 2-sided [0.096 to 0.607] — Risk difference=Response rate of spesolimab - response rate of placebo

9. Secondary Outcome: Proportion of Patients With a Generalized Pustular Psoriasis Area and Severity Index (GPPASI) 50 at Week 4
Description: Generalized Pustular Psoriasis Area and Severity Index (GPPASI) provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs).
  A higher score indicates a worse disease state, while a score of 0 indicates no disease. GPPASI 50 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 50 % reduction.
  Proportion of patients with GPPASI 50 at Week 4 is reported.
Time Frame: At Week 4.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.111 [0.031 to 0.328] | 0.543 [0.382 to 0.695]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; Confidence intervals (95%) around the risk difference were produced using the Chan and Zhang method; Test type: Other; Risk Difference (RD) = 0.432, 95% CI 2-sided [0.096 to 0.636] — Risk difference=Response rate of spesolimab - response rate of placebo

10. Secondary Outcome: Percent Change in Generalized Pustular Psoriasis Area and Severity Index (GPPASI) From Baseline at Week 4
Description: GPPASI provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 (no disease) to 72 (worse disease state). It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs).
  %GPPASI change from baseline=(GPPASI at Week 4-GPPASI at baseline) *100/(GPPASI at baseline).
  Death, any use of escape medication, OL Spesolimab at Day 8, or rescue medication with Spesolimab after Day 8, prior to observing the endpoint was considered to reflect a failure to achieve the endpoint outcome, i.e. non-response (NR).NR is not a missing value but the worst possible outcome of the endpoint. For example, if the achieved data is (NR, NR, NR, NR, NR, NR, 2, 3, 3, 3, 5) then Q1 is NR, median is NR and Q3 is 3. Planned statistical analysis were not performed due to lack of valid data.
Time Frame: Baseline and at Week 4.
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage change
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Percentage change | NA [NA to NA] — NA = "non-response", the worst possible outcome. | -60.50 [-88.37 to NA] — NA = "non-response", the worst possible outcome.

11. Secondary Outcome: Proportion of Patients With a Generalized Pustular Psoriasis Area and Severity Index (GPPASI) 50 at Week 1
Description: Generalized Pustular Psoriasis Area and Severity Index (GPPASI) provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs).
  A higher score indicates a worse disease state, while a score of 0 indicates no disease. GPPASI 50 is based on the percent reduction from baseline, generally summarized as a dichotomous outcome based on achieving over an 50 % reduction.
  Proportion of patients with GPPASI 50 at Week 1 is reported.
Time Frame: At Week 1.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Proportion of participants | 0.278 [0.125 to 0.509] | 0.429 [0.280 to 0.591]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; Confidence intervals (95%) around the risk difference were produced using the Chan and Zhang method; Test type: Other; Risk Difference (RD) = 0.151, 95% CI 2-sided [-0.138 to 0.401] — Risk difference=Response rate of spesolimab - response rate of placebo

12. Secondary Outcome: Percent Change in Generalized Pustular Psoriasis Area and Severity Index (GPPASI) From Baseline at Week 1
Description: Generalized Pustular Psoriasis Area and Severity Index (GPPASI) provides a numeric scoring for a patient's overall Generalized Pustular Psoriasis (GPP) disease state, ranging from 0 to 72. It is a linear combination of percent of surface area of skin affected by erythema, pustules, and scaling and the severity of erythema, pustules, and scaling (desquamation) over 4 body regions (head, trunk, upper limbs and lower limbs).
  A higher score indicates a worse disease state, while a score of 0 indicates no disease.
  The percent change from baseline at Week 1 is calculated as:
  % GPPASI change from baseline = (GPPASI at Week 1 - GPPASI at baseline) *100/GPPASI at baseline. If % GPPASI change from baseline is positive, it means the disease is becoming worse.
Time Frame: At Week 1.
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percentage change
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Percentage change | 1.02 [-60.47 to 36.68] | -42.80 [-69.84 to 9.49]
Statistical Analysis 1: Comparison: Placebo vs Spesolimab 900 mg i.v SD; Any assessments after death, the use of escape medication (before or after Day 8), open label spesolimab on Day 8, or rescue medication with spesolimab after Day 8 and assigned with the worst possible outcomes in rank analysis. Missing data at Week 4 were imputed and handled via assessment of ranks; Test type: Other; Median Difference (Final Values) = -16.88, 95% CI 2-sided [-67.32 to 12.76] — Median difference was calculated by modified Hodges-Lehmann method

13. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs) up to Week 1
Description: TEAEs were all Adverse Events (AEs) occurring between start of treatment and Day 8 (Day 8 excluded). AEs that started before first drug intake and deteriorated under treatment were also considered as 'treatment-emergent'.
  The exposure-adjusted incidence rate was calculated as:
  Incidence rate [1/100 patients-years] = 100 × number of patients with AE / Total AE specific time at risk [patient-years] where: Time at risk [patient-years] = (date of onset of TEAE - study drug start date + 1) /365.25
Time Frame: From start of treatment until Day 7, up to 7 days.
Population: Safety Analysis set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug on Day 1. Patients were analyzed according to the actual treatment received.
Measure: Number; unit: events per 100 patient-years at risk
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
events per 100 patient-years at risk | 6445.6 | 8650.7

14. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs) up to Week 1
Description: TEAEs were all Adverse Events (AEs) occurring between start of treatment and Day 8 (Day 8 excluded). AEs that started before first drug intake and deteriorated under treatment were also considered as 'treatment-emergent'.
Time Frame: From start of treatment until Day 7, up to 7 days.
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Participants | 12 | 27

15. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs) Within the Treatment Phase
Description: TEAEs were all Adverse Events (AEs) occurring between start of treatment and end of the residual effect period (REP) (16 weeks). AEs that started before first drug intake and deteriorated under treatment were also considered as 'treatment-emergent'.
  The exposure-adjusted incidence rate was calculated as:
  Incidence rate [1/100 patients-years] = 100 × number of patients with AE / Total AE specific time at risk [patient-years] where Time at risk where: Time at risk [patient-years] = (date of onset of TEAE - study drug start date + 1) /365.25 If, for a patient, the selected TEAE did not occur then the time at risk was censored at min
  * Date of death
  * For patients who did not roll over into the Open Label Extension (OLE) study: last contact date Visit14/15
  * For patients who rolled over into the OLE study: the 1st dose in the OLE study
  * Drug stop date + 112 days
  * Date of Day 8 if OL spesolimab was given
  * Date of rescue medication if spesolimab was given.
Time Frame: From start of treatment until end of the residual effect period (REP) but censored at any use of open label spesolimab, up to 16 weeks.
Population: as for outcome 13
Measure: Number; unit: events per 100 patient-years at risk
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
events per 100 patient-years at risk | 3083.3 | 2391.0

16. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs) Within the Treatment Phase
Description: TEAEs were all Adverse Events (AEs) occurring between start of treatment and end of the residual effect period (REP) (16 weeks). AEs that started before first drug intake and deteriorated under treatment were also considered as 'treatment-emergent'.
Time Frame: as for outcome 15
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Spesolimab 900 mg i.v SD
Number analyzed (Participants) | 18 | 35
Participants | 13 | 29

ADVERSE EVENTS:
Time Frame: Placebo and Spesolimab 900 mg i.v. SD arms: From the start of infusion of randomized medication at Day 1 (D1) of Week 1 (Wk1) until the end of its REP (16 weeks) but were censored at any use of open-label (OL) spesolimab. OL Spesolimab: From the start of OL spesolimab at Wk1/D8 until the end of its REP (16 weeks) but were censored at any use of rescue medication with spesolimab. Rescue Spesolimab: From the start of rescue medication with spesolimab until the end of its REP (16 weeks).
Description: Safety Analysis set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug on Day 1.
Groups:
- Spesolimab 900 mg i.v. SD: Patients received intravenously (i.v.) a single dose of solution for infusion containing 900 milligram (mg) of spesolimab on Day 1 (D1) of Week 1 (Wk1). Based on the subsequent treatment response, participants were then to be followed up for 12 to 28 weeks.
  If the severity and progression of the disease worsened within the first week the investigator could treat the patient with a Standard of Care (SoC) treatment of his/her choice (escape medication). If the disease condition was stable, it was recommended to wait until the primary endpoint visit (Wk1/D8) before prescribing an escape medication (SoC) since there was an option to administer open label (OL) spesolimab instead at this time. If escape medication was administered within the first week, the patient was not eligible to receive treatment with a single OL i.v. dose of 900 mg spesolimab on D8.
  If the condition of the patient worsened after Wk1/D8 patients were eligible to receive rescue treatment with open label spesolimab (only one single rescue i.v. dose of 900 mg spesolimab) after Wk1 to Wk 12.
- Open Label (OL) D8 Spesolimab 900 mg i.v.: This arm included patients who in addition to the randomized treatment (either intravenously (i.v.) placebo solution to spesolimab at Day 1 or 900 milligram (mg) i.v. spesolimab at Day 1) received also Open Label Treatment with 900 mg I.V spesolimab at Week 1 (Wk1)/Day 8 (D8).
- Rescue Spesolimab 900 mg i.v.: This arm included patients who in addition to the randomized treatment (either intravenously (i.v.) placebo solution to spesolimab at Day 1 or 900 milligram (mg) i.v spesolimab at Day 1) also one single rescue i.v. dose of 900 mg spesolimab between Week 1(Wk 1) to Week 12 (Wk 12).
Arm/Group | Placebo | Spesolimab 900 mg i.v. SD | Open Label (OL) D8 Spesolimab 900 mg i.v. | Rescue Spesolimab 900 mg i.v.
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/35 | 0/27 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/18 | 6/35 | 6/27 | 2/6
Other Adverse Events (participants affected / at risk) | 13/18 | 23/35 | 14/27 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Spesolimab 900 mg i.v. SD (N=35) | Open Label (OL) D8 Spesolimab 900 mg i.v. (N=27) | Rescue Spesolimab 900 mg i.v. (N=6)
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 3 | 4 | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | Spesolimab 900 mg i.v. SD (N=35) | Open Label (OL) D8 Spesolimab 900 mg i.v. (N=27) | Rescue Spesolimab 900 mg i.v. (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Erythropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Asthenia (General disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 4 | 2 | 2 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 2 | 0
Pustule (Infections and infestations) | 0 | 1 | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Eosinophil percentage increased (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0 | 0
High density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 1 | 1 | 0 | 0
Protein total decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 4 | 17 | 5 | 2
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the trial design, a large proportion of patients had received escape medication or non-randomized spesolimab by Week 4, based on worsening, insufficient response, or non-response. This should be taken into account for the interpretation of the results at Week 4. A large proportion of patients in both arms had been treated as non-responders at Week 4, and the true efficacy outcomes for the randomized treatment at this time-point were never observed for the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03782792/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03782792/SAP_001.pdf